CLINICAL TRIAL: NCT06692101
Title: Strategic Oral Care and Intervention for Enhanced Outcomes in Acute Ischemic Stroke Patients with Dysphagia: a Pilot Randomized Controlled Study
Brief Title: Oral Care Strategies for Stroke Patients with Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N202108021; 111HHC-02 (Other Grant/Funding Number: Taipei Medical University- Shuang Ho Hospital)
Record Dates: First submitted 2024-11-12; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2021-11

CONDITIONS: Acute Ischemic Stroke (AIS); Stroke-Associated Pneumonia (SAP); Dysphagia Following Cerebrovascular Accident
Keywords: oral care.; transcutaneous neuromuscular electrical stimulation; stroke-associated pneumonia; acute cerebral infarction; dysphagia
MeSH Terms: conditions — Ischemic Stroke; Deglutition Disorders | interventions — Dental Care Team

STUDY DESIGN:
Intervention Model Description: Study Model Description: This study is a parallel-group randomized controlled trial (RCT) employing a superiority trial design to evaluate the efficacy of combining neuromuscular electrical stimulation (NMES) with oral care compared to oral care alone and standard care in improving swallowing function and reducing the incidence of stroke-associated pneumonia (SAP) in patients with acute ischemic stroke (AIS).
  Randomization and Blinding: Participants were randomly assigned to one of the three intervention groups (Group A, Group B, or Group C) using a computer-generated randomization sequence to ensure unbiased group allocation.
  Intervention Overview:
  Group A (Oral Care Group): Focused on comprehensive oral hygiene practices administered twice daily for at least five days.
  Group B (Oral Care + NMES Group, O-NMES): Received the same oral care regimen as Group A, followed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Oral Care) (Active Comparator): Participants received oral care twice daily for at least five days. Oral care procedures included:
  * Preparation: Necessary tools and suction devices were prepared, and patients were assisted in upright sitting before oral care.
  * Oral Assessment: A flashlight and toothbrush were used to perform an oral assessment and remove food debris. Saliva was aspirated if necessary.
  * Oral Cleaning: Oral cleaning tools, including a toothbrush, dental floss, and interdental brush, were utilized with fluoridated toothpaste (fluoride >1,000 ppm, <0.5 cm³). The Bass method of brushing was employed for toothbrushing.
  * Tongue Cleaning: The anterior two-thirds of the tongue was cleaned with a moistened toothbrush following brushing.
  Interventions: Other: oral care
- Group B (O-NMES) (Active Comparator): Participants received the same oral care as Group A, and NMES therapy was administered after each oral care session. NMES therapy involved:
  * Equipment: NMES was administered using VitalStim® (Chattanooga, TN, USA).
  * Preparation: Participants were instructed to shave facial hair and cleanse the neck skin with alcohol wipes before electrode placement.
  * Electrode Placement: Four electrode pads were placed horizontally above and below the hyoid bone. (Figure 1.)
  * Stimulation Parameters: The NMES unit provided dual-pole stimulation across four channels at a fixed pulse rate of 80 Hz and a fixed biphasic pulse duration of 300 μs.
  * Session Duration and Intensity: Each session lasted 30 minutes, with the stimulation intensity gradually increased in intervals of 0.5 mA, adjusted based on patient feedback, and set to the maximum tolerance level defined by the patient.
  Interventions: Other: oral care; Device: Neuromuscular Electrical Stimulation (NMES)
- Group C (Control) (No Intervention): Participants received standard care per the unit's existing protocol, which included oral care administered by nurses and verbal education provided to patients and their caregivers to encourage oral hygiene practices at least once daily.

INTERVENTIONS:
Other: oral care — We prepared the necessary tools and suction devices, then helped patients sit upright before starting oral care. Using a flashlight and toothbrush, we assessed the mouth and removed any food debris, aspirating saliva if needed. We cleaned the teeth using a toothbrush, dental floss, and an interdental brush with a small amount of fluoridated toothpaste. The Bass method was used for brushing. Finally, we cleaned the front two-thirds of the tongue with a damp toothbrush.
  Arms: Group A (Oral Care); Group B (O-NMES)
Device: Neuromuscular Electrical Stimulation (NMES) — We used the VitalStim® device to deliver neuromuscular electrical stimulation (NMES). Before placing the electrodes, participants were asked to shave any facial hair and clean their neck skin with alcohol wipes. We positioned four electrode pads horizontally, above and below the hyoid bone. The device provided stimulation at a pulse rate of 80 Hz with a biphasic pulse duration of 300 microseconds. Each session lasted 30 minutes, with the intensity gradually increased in 0.5 mA intervals, based on the patient's comfort level, and adjusted to their maximum tolerance.
  Other Names: oral care
  Arms: Group B (O-NMES)

SUMMARY:
This study aims to evaluate whether combining neuromuscular electrical stimulation (NMES) with oral care can improve swallowing function in patients who have experienced an acute stroke and are dealing with dysphagia (difficulty swallowing). The researchers are exploring two main questions: Is this combined approach practical and manageable for patients and caregivers to use during the early stages of stroke recovery? And does this combination lead to better swallowing function and fewer stroke-related complications compared to using only oral care or traditional routine care? The goal is to identify effective strategies to support safer and faster recovery in stroke patients with swallowing difficulties.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) investigates the potential benefits of combining neuromuscular electrical stimulation (NMES) with standard oral care to improve swallowing function and reduce the incidence of stroke-associated pneumonia (SAP) in acute ischemic stroke (AIS) patients. Our study uses a rigorous, evidence-based approach to determine the clinical efficacy and feasibility of this therapeutic regimen during the critical early phase following a stroke.

Study Design

Conducted at a medical center from November 2021 to May 2023, this study enrolled AIS patients meeting specific criteria, such as being 20 years or older, diagnosed with acute ischemic stroke within 48 hours, and presenting with difficulty swallowing. Patients were randomly assigned to one of three groups:

Group A (Oral Care Group): Received comprehensive oral care twice daily for at least five days.

Group B (O-NMES Group): Received oral care paired with NMES therapy administered after each session.

Group C (Control Group): Received standard care, including routine oral hygiene practices.

Participant Screening and Baseline Assessment Upon admission, all participants underwent brain imaging (CT or MRI) to confirm stroke and exclude other conditions. Demographic data (age, gender, and cerebrovascular risk factors) and baseline assessments, such as the National Institutes of Health Stroke Scale (NIHSS) for stroke severity, were collected. Laboratory tests were performed to evaluate blood cell counts, creatinine, albumin, and glycated hemoglobin (HbA1c) levels. Participants' swallowing function and the need for nasogastric tube (NGT) insertion were also recorded.

Intervention Protocols Oral Care Procedures (Group A & B): Included the use of a toothbrush, dental floss, and fluoridated toothpaste, with the Bass method for brushing. Tongue cleaning and saliva aspiration were also performed to maintain oral hygiene.

NMES Therapy (Group B Only): NMES was delivered using the VitalStim® system. Four electrode pads were placed on the neck, and stimulation parameters were adjusted based on patient tolerance. Each NMES session lasted 30 minutes, following strict preparation and placement protocols.

Data Collection and Outcome Measures Data were collected at baseline, on day 4 (T1), and on day 8 (T2) post-stroke. Key outcomes included changes in swallowing function, assessed using tools like the Gugging Swallowing Screen (GUSS) and the incidence of SAP. The study's primary hypothesis is that combining NMES with oral care will yield better outcomes in swallowing function and reduce pneumonia risk compared to oral care alone or standard care.

Assessment Tools NIHSS: Used to evaluate stroke severity, focusing on items like facial palsy, language, and speech that may influence oral and swallowing control.

ROAG: Assesses oral health status across multiple categories, with higher scores indicating more severe oral health issues.

GUSS: A comprehensive tool to screen and monitor swallowing function, facilitating the identification of impairments and personalized care.

Study Implications This research is designed to contribute valuable insights into stroke rehabilitation and offer evidence-based guidelines for enhancing clinical care. By exploring different treatment strategies, we aim to inform future practices in managing dysphagia and preventing SAP in stroke patients, ultimately improving recovery outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years.
2. First diagnosis of acute ischemic stroke (AIS) and hospitalization.
3. Stroke onset within 48 hours.
4. NIHSS score ≥ 5 upon admission, with at least one of the following NIHSS items: facial palsy, language, or dysarthria.
5. Difficulty swallowing upon admission, indicated by a Gugging Swallowing Screen-Indirect Test score < 5.
6. Ability to communicate verbally or in writing and provide informed consent.

Exclusion Criteria:

1. Diagnosed with pneumonia or exhibiting clinical symptoms of infection upon admission.
2. Requiring mechanical ventilation.
3. Use of antibiotics or immunosuppressants within the past month.
4. Eligible for intravenous recombinant tissue plasminogen activator (r-tPA) or mechanical thrombectomy.
5. History of seizure or epilepsy.
6. Severe communication impairment due to cognitive deficits or psychological disorders.
7. Presence of oral-pharyngeal tumors or a history of extensive surgery or radiotherapy in the head and neck region.
8. Use of electrically sensitive biomedical devices (e.g., defibrillators or pacemakers).
9. Pregnancy.

Min Age: 20 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Changes in stroke severity and swallowing function (GUSS) at three-time points-baseline (T0), the fourth-day post-stroke (T1), and the eighth-day post-stroke (T2) | From enrollment to the end of treatment at day 8 post-stroke. Outcome measures were assessed at baseline (day 0), day 4, and day 8 post-stroke.
  The Revised Oral Assessment Guide (ROAG) is a standardized tool for comprehensive oral health status and function assessment. It comprises eight categories: voice, lips, mucous membranes, tongue, gums, teeth or dentures, saliva production, and swallowing function. Assessors describe each category and rate them on a scoring scale, where one indicates healthy, 2 indicates minor problems, and 3 indicates severe problems. The ROAG total score ranges from 3 to 24 points, with higher scores suggesting the need for more care and attention to the participant's oral health.
Changes in stroke severity and swallowing function (ROAG) at three-time points-baseline (T0), the fourth-day post-stroke (T1), and the eighth-day post-stroke (T2) | From enrollment to the end of treatment at day 8 post-stroke. Outcome measures were assessed at baseline (day 0), day 4, and day 8 post-stroke.
  The Bedside Gugging Swallow Screen (GUSS) is a screening tool used to assess swallowing function, aiming to comprehensively evaluate a patient's ability to swallow at different viscosities. It utilizes a scoring system ranging from 0-20 points, with higher scores indicating better swallowing function. GUSS consists of a preliminary assessment, the Indirect Swallow Test (5 points), and the Direct Swallow Test (15 points). The first part includes a simple saliva swallow test, observing the patient's alertness, voluntary cough, throat clearing, and saliva swallowing. The second part comprises three subtests challenging the patient's ability to swallow semi-solids, liquids, and solids. This graded assessment design allows for a detailed evaluation of different viscosities, aiding in the timely detection of swallowing impairments and facilitating personalized dietary recommendations.
Changes in stroke severity and swallowing function (NIHSS) at three-time points-baseline (T0), the fourth-day post-stroke (T1), and the eighth-day post-stroke (T2) | From enrollment to the end of treatment at day 8 post-stroke. Outcome measures were assessed at baseline (day 0), day 4, and day 8 post-stroke.
  The National Institutes of Health Stroke Scale (NIHSS) comprises 15 neurological examination items and is commonly used to assess stroke severity. Due to its simplicity, repeatability, reliability, and validity, NIHSS scores have become a widely utilized indicator in stroke models for evaluating Acute Ischemic Stroke (AIS) outcomes. Although the NIHSS scale does not directly assess swallowing function, language impairments or speech difficulties may affect oral control in patients, potentially correlating with swallowing function to some extent. Similarly, facial palsy is associated with control of facial and oral muscles, thereby impacting swallowing function. In this study, we included patients with at least one of the NIHSS subitems involving facial palsy, language impairment, or speech difficulty to thoroughly evaluate the treatment effects and the risk of post-stroke pneumonia in AIS patients exhibiting these symptoms.
Reducing stroke-associated pneumonia (SAP) incidence in acute stroke patients | Comparison of SAP occurrence within seven days after stroke.
  In 2014, a consensus meeting was held in Manchester, UK, and after literature search, evidence review and consensus negotiation, SAP was defined as respiratory infection within seven days after stroke. SAP diagnosis is mainly based on the diagnostic criteria for pneumonia proposed by the Centers for Disease Control and Prevention (CDC): typical pulmonary symptoms (tachypnea, inspiratory crackles, bronchial breathing) or chest X-ray Abnormalities (infiltrates, parenchymal lesions) and other evidence such as fever (temperature >38°C), cough with purulent sputum, or isolation of pathogens by blood/sputum culture (Garner et al., 1988).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Shuang Ho Hospital, Taipei Medical University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The content is not yet complete.